CLINICAL TRIAL: NCT03464461
Title: Dosing of Ketorolac for Four Classes of Complaints in the Emergency Department
Brief Title: Dosing of Ketorolac in the Emergency Department
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Pandemic related supply shortages and slowed enrollment.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Matthew Robinson, Associate Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010856
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Results first posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain | interventions — Ketorolac

STUDY DESIGN:
Intervention Model Description: 4 groups with 3 different treatments
Who Masked: Participant, Care Provider
Masking Description: blinded drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 0 mg (Placebo Comparator): 0 mg ketorolac - placebo
  Interventions: Drug: Ketorolac
- 10 mg (Active Comparator): 10 mg ketorolac - low dose ketorolac
  Interventions: Drug: Ketorolac
- 30 mg (Active Comparator): 30 mg ketorolac - usual dose ketorolac
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — IV drug
  Other Names: Use of placebo, low, usual dose ketorolac

SUMMARY:
The optimal dose of ketorolac in the Emergency Department setting is no clear. We will compare 3 doses to determine the optimal dose.

DETAILED DESCRIPTION:
Patients from 4 groups will be treated with 3 different doses of ketorolac. The groups are 1. headache 2. abdominal pain 3. musculo-skeletal pain 4. viral syndrome. The doses will be 0, 10, 30mgs of ketorolac to clarify the placebo effect and the optimal dosage as a function of condition.

ELIGIBILITY:
Inclusion Criteria:

> 18 y/o

Exclusion Criteria:

pregnant allergic other contraindication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Robinson, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Health Care, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were excluded if they were giving medications that could interfere with study results, if study medication could not be administered, at the providers discretion, or if the participant decided to withdraw from the study.
  31 participants signed consent but withdrew/were excluded before study drug administration 4 participants were excluded after study drug administration (see below)
Period: Overall Study
Arm/Group | 0 mg | 10 mg | 30 mg
Started | 83 | 92 | 83
Completed | 82 | 89 | 83
Not Completed | 1 | 3 | 0
Not completed — exclusionary medication given , | 1 | 2 | 0
Not completed — Physician Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 mg | 10 mg | 30 mg | Total
Number analyzed (Participants) | 82 | 89 | 83 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (17) | 44 (16) | 41 (16) | 43 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 51 | 46 | 128
  Male | 51 | 38 | 37 | 126
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 82 | 89 | 83 | 254
Baseline Pain Score [Mean (Standard Deviation); unit: millimeters (mm)] — The average number of millimeters measured from the 0mm end of the 100mm long Visual Analog Scale (VAS) line to the mark on the line made by the participants indicating their pain level before given the study treatment.
  millimeters (mm) | 67.2 (15.1) | 65.3 (15.6) | 66.4 (16.7) | 66.30 (21.39)

OUTCOME MEASURES:

1. Primary Outcome: Difference of Pain Intensity Before and 30 Minute After Study Drug Administration in Participants With Any Pain Type
Description: The outcome measure is the average change in pain score.
  Change in pain score is calculated for each participant by subtracting the post-treatment pain score from the pretreatment pain score (i.e. pre-treatment pain score minus post-treatment pain score), then averaging them within each group.
  The pain score is collected using the visual analog scale, which is a 100mm line that participants make a mark on to indicate their pain intensity. The line is then measured from the left end of the line to where the mark was made. The minimum value is 0mm (left end of the line) being no pain and the maximum value is 100mm (right end of the line) being the worst pain possible.
Time Frame: 30 minutes
Population: Patients presenting to the Emergency Department with pain that falls in one of the for categories: abdominal, headache, trauma/musculoskeletal, viral
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0 mg | 10 mg | 30 mg
Number analyzed (Participants) | 82 | 89 | 83
mm | 15.1 (18.5) | 15.6 (19.4) | 16.7 (20.7)
Statistical Analysis 1: Comparison: 0 mg vs 10 mg vs 30 mg; Test type: Other — non-parametric; p = 0.9844, Kruskal-Wallis

2. Primary Outcome: Difference of Pain Intensity Before and 30 Minute After Study Drug Administration in Participants With Abdominal Pain
Description: as for outcome 1
Time Frame: 30 minutes
Population: Patients presenting to the Emergency Department with abdominal pain
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0 mg | 10 mg | 30 mg
Number analyzed (Participants) | 37 | 46 | 47
mm | 12.4 (16.5) | 19.4 (19.9) | 22.1 (21.0)
Statistical Analysis 1: Comparison: 0 mg vs 10 mg vs 30 mg; Test type: Other — non-parametric; p = 0.1580, Kruskal-Wallis

3. Primary Outcome: Difference of Pain Intensity Before and 30 Minute After Study Drug Administration in Participants With Headache
Description: as for outcome 1
Time Frame: 30 minutes
Population: Patients presenting to the Emergency Department with headache
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0 mg | 10 mg | 30 mg
Number analyzed (Participants) | 9 | 4 | 7
mm | 13.3 (14.8) | 10.8 (8.7) | 11.1 (18.4)
Statistical Analysis 1: Comparison: 0 mg vs 10 mg vs 30 mg; Test type: Other — non-parametric; p = 0.8730, Kruskal-Wallis

4. Primary Outcome: Difference of Pain Intensity Before and 30 Minute After Study Drug Administration in Participants With Trauma/Musculoskeletal Pain
Description: as for outcome 1
Time Frame: 30 min
Population: Patients presenting to the Emergency Department with trauma/musculoskeletal pain
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0 mg | 10 mg | 30 mg
Number analyzed (Participants) | 24 | 27 | 19
mm | 16.5 (21.0) | 5.4 (15.6) | 10.0 (19.0)
Statistical Analysis 1: Comparison: 0 mg vs 10 mg vs 30 mg; Test type: Other — non-parametric; p = 0.0740, Kruskal-Wallis

5. Primary Outcome: Difference of Pain Intensity Before and 30 Minute After Study Drug Administration in Participants With Viral Pain
Description: as for outcome 1
Time Frame: 30 min
Population: Patients presenting to the Emergency Department with viral pain
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 0 mg | 10 mg | 30 mg
Number analyzed (Participants) | 12 | 12 | 10
mm | 21.8 (19.3) | 25.4 (17.5) | 8.4 (15.7)
Statistical Analysis 1: Comparison: 0 mg vs 10 mg vs 30 mg; Test type: Other — non-parametric; p = 0.0984, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Approximately 40 minutes, from the time of consent until post-treatment pain score was obtained
Arm/Group | 0 mg | 10 mg | 30 mg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/89 | 0/83
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/89 | 0/83
Other Adverse Events (participants affected / at risk) | 0/82 | 0/89 | 0/83

LIMITATIONS AND CAVEATS:
Study enrollment ended early, resulting in less than half of the number of participants needed according to the power analysis. Our study site was closed to enrollment during the recent pandemic, and there was major supply chain issues for saline and IV equipment. Ultimately the study was closed due to the extenuating circumstances.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT03464461/Prot_SAP_002.pdf
  • Informed Consent Form (2022-03-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT03464461/ICF_001.pdf